CLINICAL TRIAL: NCT00136747
Title: Developing Medication For Tobacco Addiction: NMDA Agents
Brief Title: The Effects of Memantine and Bupropion on Acute, Reinforcing, and Conditioned Effects of Cigarettes - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #4725(1); R01DA017572 (NIH); R01DA017572-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco use
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use | interventions — Memantine; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- BUPROPION (Experimental): Participants receive 20 mg bid of memantine, placebo, or bupropion in a double-blind crossover design and are maintained on active or placebo medication for 5 or 10 days before the inpatient testing
  Interventions: Drug: bupropion
- placebo (Experimental): Participants receive 20 mg bid of memantine, placebo, or bupropion in a double-blind crossover design and are maintained on active or placebo medication for 5 or 10 days before the inpatient testing
  Interventions: Drug: placebo
- memantine (Experimental): Participants receive 20 mg bid of memantine, placebo, or bupropion in a double-blind crossover design and are maintained on active or placebo medication for 5 or 10 days before the inpatient testing
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Two capsules of Memantine twice daily for 12 days.
  Arms: memantine
Drug: bupropion
  Arms: BUPROPION
Drug: placebo
  Arms: placebo

SUMMARY:
One of nicotine's effects on the body is at the level of the NMDA receptors in the brain. Memantine is a drug that also affects NMDA receptors, making it a candidate for the treatment of nicotine addiction. The purpose of this study is to evaluate the effectiveness of memantine using a laboratory model of tobacco addiction. The investigators will compare the effects of memantine with bupropion, medication currently used to facilitate smoking cessation.

DETAILED DESCRIPTION:
Tobacco use is the leading preventable cause of death in the United States. Recent research on the effects of nicotine on the brain and behavior presents an opportunity to advance medication development. Neurotransmission at NMDA receptors in the brain is associated with learning and memory and has been linked to many of nicotine's effects on humans. It is possible that altering NMDA neurotransmission may be helpful in treating nicotine addiction.

The goal of this study is to develop a laboratory model for early-stage testing of new and existing compounds for the treatment of tobacco and nicotine addiction. Specifically, the study will assess the effect of memantine, a non-competitive NMDA antagonist, versus bupropion, a medication currently used to facilitate smoking cessation, on various behavioral aspects related to smoking behavior, including reinforcement and cue-reactivity.

This double-blind, randomized assignment study will consist of three distinct phases (placebo, bupropion, and memantine). Each phase will include 10 days of outpatient medication maintenance, followed by 3 days of inpatient testing. During the outpatient phase, study visits will occur every 2 to 3 days. At these visits, compliance and side effects of medication will be monitored, smoking diaries will be collected, and medication will be dispensed. During the inpatient period participants will be allowed to smoke only at designated times. A variety of assessment will be conducted, including abstinence symptoms, acute effects of cigarettes, responses to cigarette cues, and cigarette self-administration.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of nicotine dependence with psychological dependence
* Smokes at least 15 cigarettes per day for the three months prior to enrollment
* Currently not seeking treatment for nicotine dependence
* Medically healthy on the basis of physical examination and medical history, vital signs, EKG, and laboratory tests
* Females must use an effective method of contraception for the duration of the study

Exclusion Criteria:

* DSM-IV diagnosis of abuse or dependence on alcohol or drugs other than nicotine
* Current Axis I diagnosis or current treatment with psychotropic medications within the three months prior to enrollment
* History of schizophrenia or other psychotic disorders, bipolar disorder, or anxiety disorders
* Currently seeking treatment for nicotine disorders
* On parole or probation
* History of seizures or head trauma with loss of consciousness, brain contusion, or fracture
* History of significant recent violent behavior
* Blood pressure greater than 150/90
* History of eating disorders
* History of allergic reaction to any of the study medications
* Pregnant

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2004-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Response to cigarette cues | Days 11-13
Smoking behavior | Days 11-13

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States